CLINICAL TRIAL: NCT07035990
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses and Multiple Ascending Doses of SION-451, and Multiple Dose Combinations of SION-451 and Complementary Modulators SION-2222 and SION-109 in Healthy Participants.
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Dose Combinations of SION-451 and Complementary Modulators SION-2222 and SION-109 in Healthy Participants.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sionna Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SION-451-101; ACTRN12624000849895 (Registry Identifier: Australian New Zealand Clinical Trials Registry); ACTRN12624000848505 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2025-06-04; First posted 2025-06-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cystic Fibrosis (CF)
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SION-451 + SION-2222 (Experimental): All participants who receive SION-451 in combination with SION-2222
  Interventions: Drug: SION-451; Drug: SION-2222
- Placebo matched to SION-451 and SION-2222 (Placebo Comparator)
  Interventions: Drug: Placebo SION-451; Drug: Placebo SION-2222
- SION 451 + SION 109 (Experimental): All participants who receive SION-451 in combination with SION-109
  Interventions: Drug: SION-451; Drug: SION-109
- Placebo matched to SION-451 and SION-109 (Placebo Comparator)
  Interventions: Drug: Placebo SION-451; Drug: Placebo SION-109

INTERVENTIONS:
Drug: SION-451 — * Pharmaceutical form: tablet
  * Route of administration: oral
  Arms: SION 451 + SION 109; SION-451 + SION-2222
Drug: SION-2222 — * Pharmaceutical form: capsule
  * Route of administration: oral
  Arms: SION-451 + SION-2222
Drug: SION-109 — * Pharmaceutical form: tablet
  * Route of administration: oral
  Arms: SION 451 + SION 109
Drug: Placebo SION-451 — Placebo matched to SION-451
  Arms: Placebo matched to SION-451 and SION-109; Placebo matched to SION-451 and SION-2222
Drug: Placebo SION-2222 — Placebo matched to SION-2222
  Arms: Placebo matched to SION-451 and SION-2222
Drug: Placebo SION-109 — Placebo matched to SION-109
  Arms: Placebo matched to SION-451 and SION-109

SUMMARY:
The purpose of Parts D and E of this Phase 1 study are to evaluate the safety, tolerability, and pharmacokinetics of multiple dose combinations of SION-451 and complementary modulators SION-2222 and SION-109 in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1 randomized, double-blind, placebo-controlled study. Parts D and E will evaluate the safety, tolerability, and pharmacokinetics of multiple dose combinations of SION-451 and complementary modulators SION-2222 and SION-109 in healthy participants. Parts A, B, and C of this study have completed dosing.

Part D will involve multiple dosing of SION-451 and SION-2222 in combination. Part E will involve multiple dosing of SION-451 and SION-109 in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adult participants aged 18 to 55 years, inclusive, at the time of consent.
2. Weight of at least 45 kg and body mass index between 18.0 and 32.0 kg/m2, inclusive, at Screening.
3. Participant is willing to abstain from alcohol, caffeine, smoking and nicotine-containing products for 72 hours prior to Day -1 through the duration of the study. Participant is willing to abstain from eating cruciferous vegetables, charcoal-grilled meats, and poppy seeds for 48 hours prior to dosing throughout the duration of the study.
4. Participant has read, understood, and voluntarily provided written informed consent
5. Participant has an understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Participant has clinically significant, in the opinion of the investigator, current or recurrent illness, such as cardiovascular (including but not limited to known structural cardiac abnormalities, family history of long QT syndrome, or cardiac syncope or recurrent, idiopathic syncope), neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality which may affect safety or clinical laboratory evaluations.
2. Participant has a history of malignancy, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of recurrence for at least 1 year.
3. Participant has clinically significant abnormalities, in the opinion of the investigator, on ECG, physical examination, or vital sign assessment at Screening or Day -1.
4. Participant has any single reading of QTcF >470 ms (females) or >450 ms (males) at Screening or Day -1.
5. Chronic or habitual alcohol (>10 standard drinks per week) or tobacco (>10 cigarettes per week) use or use of recreational drugs (>1 use per month). The Investigator may exclude a participant with lower levels of alcohol, tobacco, or recreational drug use based on discretion and the pattern or history of use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of treatment emergent adverse events [Safety and Tolerability] of SION-451 and SION-109 when administered in combination to healthy participants | From Day 1 through day 21
  Adverse reactions to the study drug combination SION-451 and SION-109 will be measured.
To evaluate the incidence of treatment emergent adverse events [Safety and Tolerability] of SION-451 and SION-2222 when administered in combination to healthy participants | From Day 1 through day 21
  Adverse events to the study drug combination SION-451 and SION-2222 will be measured

SECONDARY OUTCOMES:
Cmax of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Tmax of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
AUC of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
t1/2 of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Volume of distribution of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Apparent total clearance of SION-451 and SION-2222 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Cmax of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Tmax of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17
AUC of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17
t1/2 of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Volume of distribution of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17
Apparent total clearance of SION-451 and SION-109 in plasma when administered in combination to healthy participants | From Day 1 through day 17

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ryan, MBBS, BMedSc, PhD, DPM, FFPM, Principal Investigator — Nucleus Network
Locations (2):
- Australia (2):
  - Nucleus Network, Brisbane, Queensland
  - Nucleus Network, Melbourne, Victoria